CLINICAL TRIAL: NCT06152250
Title: Characterization of the Intrahepatic Inflammatory Microenvironment in Patients With Non-alcoholic Steatohepatitis by Transcriptomics, Immunophenotyping and Functional Proteomics: Profil-NASH
Brief Title: Characterization of the Intrahepatic Inflammatory Microenvironment in Patients With Non-alcoholic Steatohepatitis
Acronym: Profil-NASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_1059
Record Dates: First submitted 2023-11-15; First posted 2023-11-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases
Keywords: intra-hepatic immune responses; liver inflammation; non-alcoholic fatty liver; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Liver Diseases; Hepatitis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Liver Fine-Needle Aspiration, blood sampling and clinical evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Fine-Needle Aspiration, blood sampling and clinical evaluation (Other): At the time of inclusion, when liver biopsy will be performed as part of routine medical management, fine-needle aspiration and blood sampling will also be made in all patients.
  The procedure will be performed in the Day Hospital, immediately after the liver biopsy and after the same local anaesthetic. Specific blood sampling will be made the same day (20mL of plasma in Ethylenediaminetetraacetic Acid Tetrasodium (EDTA) tubes and 20 mL of plasma in heparin tubes).
  Clinical information will be collected in electronic Case Report Form (e-CRF). After the procedure, the patient will be monitored as part of the usual protocol. No follow-up data are expected with Profile-NASH.
  Interventions: Other: Liver Fine-Needle Aspiration

INTERVENTIONS:
Other: Liver Fine-Needle Aspiration — At the time of inclusion, when liver biopsy will be performed as part of routine medical management, fine-needle aspiration will also be made in all patients.
  The procedure will be performed in the Day Hospital, immediately after the liver biopsy.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a nosological entity that groups together non-alcoholic fatty liver (NAFL) and non-alcoholic steatohepatitis (NASH). Unlike NAFL, NASH is characterized by intrahepatic inflammation, and is solely at risk of progression to cirrhosis and hepatocellular carcinoma (HCC).

It is currently estimated that NAFLD affects approximately 25% of the world's adult population, and its incidence is rising in all regions of the world. Nevertheless, of all patients with NAFLD, only ~25% have NASH.

Identifying patients with NASH is therefore crucial, determining the need for follow-up to detect the onset of fibrosis and/or HCC, and eventual access to therapeutic trials. Furthermore, intrahepatic inflammation, the initial driver of NASH, appears to play an important role in the development of fibrosis and HCC, which can occur in the absence of cirrhosis in these patients. However, few studies have been carried out in humans to date, with data mainly coming from mouse models.

An innovative technique, Fine-Needle Aspiration (FNA), enables to obtain cells from the liver compartment, including large numbers of immune cells. In participants with NAFLD and indication of liver biopsy, a FNA will also be performed. Forty patients will be included, with ~75% of NASH and ~25% of NAFL expected. The investigators will study the phenotypic and functional characteristics of human intrahepatic inflammatory cells obtained by the FNA with different innovative techniques (RNAseq, multiparameter immunophenotyping, single-cell secretome and phosphoproteome). Peripheral Blood Mononuclear Cells and circulating microRNAs, known to regulate immune responses, will also be analysed.

The hypothesis of Profile-NASH is that intrahepatic inflammatory profiles differ between NASH and NAFL, and is associated with fibrosis progression and carcinogenesis.

This pilot study, based on high-definition technologies, will provide precise new insights into the quality of intrahepatic inflammation and the mechanisms favoring the transition from NAFL to NASH and its progression. Precise analysis of the intrahepatic inflammatory microenvironment will enable the investigators to identify new players in the pathogenesis of NASH, and potential future therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* patient with a clinical diagnosis of NAFLD: steatosis detected on imaging and exclusion of secondary causes of steatosis (drugs, genetics, alcohol consumption >30 g/d in men and 20 g/d in women, chronic viral infection), in the absence or presence of an associated metabolic syndrome
* and with significant liver fibrosis (≥ F2) on at least one non-invasive test (FibroScan®, Fibrometer®, NAFLD Fibrosis Score);
* Patient of legal age (age ≥ 18 years);
* Patient willing to undergo liver biopsy ;
* Patient consenting to inclusion in the study after being informed and obtaining written consent;
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Decompensated cirrhosis or clinically significant portal hypertension (clinical, radiological or endoscopic signs of portal hypertension; presence of hepatocellular insufficiency);
* Secondary causes of steatosis, including chronic viral hepatitis, drugs, excessive alcohol consumption according to World Health Organization (WHO) criteria (> 30 g/d in men and 20 g/d in women), genetic mutations;
* Any other cause of liver disease: genetic hemochromatosis, autoimmune liver disease, etc. (non-exhaustive list);
* Presence of HCC at the time of inclusion;
* Contraindications to liver biopsy (identical to those for FNA): coagulation disorders, biliary tract dilatation, intrahepatic tumor;
* Pregnant, parturient or breast-feeding women;
* Persons deprived of their liberty by judicial or administrative decision;
* adults under legal protection (guardianship, curators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-29 (Actual); Primary Completion 2029-01-29 (Estimated); Study Completion 2029-01-29 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the comparison of transcriptomic profiles between NAFL and NASH patients. | At the time of the procedure liver biopsy at Day 1
  Cells collected from the RNA extraction plasma cell will be analyzed with technique:
  - Transcriptomic analysis (RNA-Seq) The data obtained by these analyses will be compared between patients with NASH vs. NAFL, using multiple testing corrections.
The primary endpoint is the secretome and single-cell phosphoproteome between NAFL and NASH patients. | At the time of the procedure liver biopsy at Day 1
  Cells collected from the FNA procedure will be analyzed with technique:
  - Single-cell secretome and phosphoproteome by ISOPLEXIS® The data obtained by these analyses will be compared between patients with NASH vs. NAFL, using multiple testing corrections.
The primary endpoint is the immunophenotyping of intrahepatic mononuclear cells between NAFL and NASH patients. | At the time of the procedure liver biopsy at Day 1
  Cells collected from the peripheral blood mononuclear cells will be analyzed with technique:
  - Multiparameter immunophenotyping by spectral cytometry The data obtained by these analyses will be compared between patients with NASH vs. NAFL, using multiple testing corrections.

SECONDARY OUTCOMES:
Comparison of transcriptome profiles between patients with significant liver fibrosis (≥ F2) and patients without significant fibrosis (F0/F1). | At the time of the procedure liver biopsy at Day 1
  This secondary outcome is a subgroup analysis of the primary outcome, only in the group " NASH ", between patients with or without significant liver fibrosis. The classification of patients according to their fibrosis stage will be made after histological evaluation of the liver biopsy.
  Cells collected from the RNA extraction plasma cell will be analyzed with technique:
  - Transcriptomic analysis (RNA-Seq)
Comparison of secretome and single-cell phosphoproteome between patients with significant liver fibrosis (≥ F2) and patients without significant fibrosis (F0/F1). | At the time of the procedure liver biopsy at Day 1
  This secondary outcome is a subgroup analysis of the primary outcome, only in the group " NASH ", between patients with or without significant liver fibrosis. The classification of patients according to their fibrosis stage will be made after histological evaluation of the liver biopsy.
  Cells collected from the FNA procedure will be analyzed with technique:
  - Single-cell secretome and phosphoproteome by ISOPLEXIS®
Comparison of the immunophenotyping profiles of intrahepatic mononuclear cells between patients with significant liver fibrosis (≥ F2) and patients without significant fibrosis (F0/F1). | At the time of the procedure liver biopsy at Day 1
  This secondary outcome is a subgroup analysis of the primary outcome, only in the group " NASH ", between patients with or without significant liver fibrosis. The classification of patients according to their fibrosis stage will be made after histological evaluation of the liver biopsy.
  Cells collected from the peripheral blood mononuclear cells will be analyzed with technique:
  - Multiparameter immunophenotyping by spectral cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Service Hepato Gastrologie, Lyon, Auvergne-Rhône-Alpes, France